CLINICAL TRIAL: NCT03362827
Title: Assessment of Long-term Potentiation (LTP)-Like Pain Amplification in Chronic Low Back Pain Patients
Brief Title: Assessment of LTP-like Pain Amplification in Chronic Low Back Pain Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Chenjun, Department of Spine Surgery, Peking University People's Hospital
Other Study IDs: BackpainLTP
Record Dates: First submitted 2017-11-25; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Low Back Pain
Keywords: Low back pain; Long-term potentiation; Hyperalgesia; Allodynia
MeSH Terms: conditions — Low Back Pain; Hyperalgesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic low back pain patients: People must have experienced low back pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.
  Interventions: Other: Chronic low back pain patients
- Subjects without chronic low back pain: Participants must not have presented episodes of low back pain for more than 7 days in the last 12 months.
  Interventions: Other: Subjects without chronic low back pain

INTERVENTIONS:
Other: Chronic low back pain patients — People must have experienced low back pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.
  Groups: Chronic low back pain patients
Other: Subjects without chronic low back pain — These participants must not have presented episodes of low back pain for more than 7 days in the last 12 months.
  Groups: Subjects without chronic low back pain

SUMMARY:
The present study is aimed to assess the LTP-like pain amplification in chronic low back pain patients to explore the central and peripheral effect for pain LTP.

DETAILED DESCRIPTION:
This study is a cross-sectional study. Two groups, including low back pain group and healthy subjects group will be arranged in this study. 50 subjects will be recruited in each group, The healthy subjects were matched for sex and age in relation to the low back pain group. Conditioning electrical stimulation (100 Hz, repeated 5 times with 10 s intervals, 500 impulses) using circular pin electrodes will be used in both groups to induce LTP-like pain amplification. The pain intensity changes to pinprick and light touch stimuli will be compared between two groups.

ELIGIBILITY:
1. Chronic low back pain patients

   Inclusion Criteria:
   * Age 21-80 years old.
   * People must have experienced low back pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.

   Exclusion Criteria:
   * Age below 21 or over 80 years old.
   * Patients were excluded if they had taken pain medications on the day of the assessment or if they had serious spinal pathologies, such as fractures, tumors or inflammatory diseases, such as ankylosing spondylitis, nerve root compromise confirmed by clinical neurological tests or severe cardiorespiratory diseases. Those who were pregnant, patients with cancer and those with a cardiac pacemaker were also excluded.
2. Healthy volunteers.

Inclusion Criteria:

* Age 21-80 years old.
* These participants must not have presented episodes of low back pain for more than 7 days in the last 12 months.

Exclusion Criteria:

* Age below 21 or over 80 years old.
* These participants have presented episodes of low back pain for more than 7 days in the last 12 months.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Chronic low back pain patients Age 21-80 years old.People must have experienced low back pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.Patients were excluded if they had taken pain medications on the day of the assessment or if they had serious spinal pathologies, such as fractures, tumors or inflammatory diseases. Those who were pregnant, patients with cancer and those with a cardiac pacemaker were also excluded.
  2. Healthy volunteers. Age 21-80 years old.These participants must not have presented episodes of low back pain for more than 7 days in the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of pain intensity to pinprick stimuli | The pinprick sensation will be measured three times before and six times after the conditioning electrical stimulation with 10 minutes interval throughout the experiment (90 minutes).
  Mechanical pinprick-evoked perception was assessed by three weighted pinprick stimulators which were randomly applied in the area adjacent to the conditioned site. The subjects indicated the perceived intensity on the same visual analogue scale(VAS).

SECONDARY OUTCOMES:
Perception Features of conditioning electrical stimulation (CES) | All subjects will rate the pain ratings during the 50 seconds stimulation.
  The subjects were asked to rate continuously the magnitude of pain induced by the 100 Hz CES using a hand-held visual analogue scale (VAS) device. These VAS ratings were sampled by a computer. The VAS ranges from "0"(no sensation") to "100" (most imaginable pain) where "30" means pain threshold.
Change of pain intensity to light-stroking stimuli | The light-touch sensation will be measured three times before and six times after the conditioning electrical stimulation with 10 minutes interval throughout the experiment (90 minutes).
  A cotton swab was used for light stroking stimuli (~100mN) for assessing the tactile perception around the conditioned site.
Change of pain intensity to single electrical stimulation (SES) | The pain ratings to SES will be measured three times before and six times after the conditioning electrical stimulation with 10 minutes interval throughout the experiment (90 minutes).
  A single rectangular 1 ms constant-current electrical stimulation was applied as a homotopic electrical test stimulus using the same conditioning electrode placed at the conditioned site.

CONTACTS AND LOCATIONS:
Overall Officials: Chenjun Liu, Ph.D., Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biurrun Manresa JA, Morch CD, Andersen OK. Long-term facilitation of nociceptive withdrawal reflexes following low-frequency conditioning electrical stimulation: a new model for central sensitization in humans. Eur J Pain. 2010 Sep;14(8):822-31. doi: 10.1016/j.ejpain.2009.12.008. Epub 2010 Jan 27. PMID 20110183
- [Background] Mouraux A, Iannetti GD, Plaghki L. Low intensity intra-epidermal electrical stimulation can activate Adelta-nociceptors selectively. Pain. 2010 Jul;150(1):199-207. doi: 10.1016/j.pain.2010.04.026. Epub 2010 May 26. PMID 20510515
- [Background] Morch CD, Hennings K, Andersen OK. Estimating nerve excitation thresholds to cutaneous electrical stimulation by finite element modeling combined with a stochastic branching nerve fiber model. Med Biol Eng Comput. 2011 Apr;49(4):385-95. doi: 10.1007/s11517-010-0725-8. Epub 2011 Jan 5. PMID 21207174
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Xia W, Morch CD, Andersen OK. Test-Retest Reliability of 10 Hz Conditioning Electrical Stimulation Inducing Long-Term Potentiation (LTP)-Like Pain Amplification in Humans. PLoS One. 2016 Aug 16;11(8):e0161117. doi: 10.1371/journal.pone.0161117. eCollection 2016. PMID 27529175